CLINICAL TRIAL: NCT01361854
Title: Comparison of 2 Different Hook-up Protocols to Perform Home-based Polysomnography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, chest physician, Centre Hospitalier Universitaire Saint Pierre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: AK/11-05-42/4024
Record Dates: First submitted 2011-05-26; First posted 2011-05-27 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Sleep Disordered-breathing
Keywords: polysomnography; portable monitoring; sleep; sleep disordered breathing; home based polysomnography
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Polysomnography

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- polysomnography for suspicion of SDB (Experimental): adults, suspects of suffering from sleep disordered-breathing, who must undergo a diagnostic polysomnography
  Interventions: Device: polysomnography

INTERVENTIONS:
Device: polysomnography — home-based polysomnography with hook-up performed ar at home or in the hospital
  Other Names: sleep study

SUMMARY:
Comparison of 2 hook-up protocols to perform home-based sleep studies in patients suspected of sleep-disordered breathing.

First one: hook-up is performed in the hospital, around 4 PM, and the patient go home with the portable monitoring.

Second one: hook-up is performed home, around 7 PM, and the patient has not to move after hook-up.

DETAILED DESCRIPTION:
All the patients will undergo 2 polysomnographies, according to two different hook-up protocols, within 2 weeks. Order of the exams will be randomized.

We hypothesised that quality of recording is better when hook-up is performed at home.

Final polysomnographic diagnosis, with the 2 different techniques, must be similar.

ELIGIBILITY:
Inclusion Criteria:

* adult,
* suspects of SDB,
* leaving home,
* at maximum 30km around the hospital

Exclusion Criteria:

* suspicion of other sleep disorders
* children

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: marie Bruyneel, MD, Principal Investigator — CHU St Pierre
Locations (1):
- CHU Saint Pierre, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Hook-up First Then Hook-up in the Hospital: adults, suspects of suffering from sleep disordered-breathing, who must undergo a diagnostic polysomnography
  polysomnography: home-based polysomnography with hook-up performed at home first.
  Croosover design. 2nd polysomnography with in-lab hook-up performed within 2 weeks
- Hospital Hook-up First, Then Home Hook-up: adults, suspects of suffering from sleep disordered-breathing, who must undergo a diagnostic polysomnography
  polysomnography: home-based polysomnography with hook-up performed at the hospital Croosover design. 2nd polysomnography with home hook-up performed within 2 weeks
Period: Day 1
Arm/Group | Home Hook-up First Then Hook-up in the Hospital | Hospital Hook-up First, Then Home Hook-up
Started | 51 | 51
Completed | 47 | 48
Not Completed | 4 | 3
Period: Wash-out, Maximum 2 Weeks
Arm/Group | Home Hook-up First Then Hook-up in the Hospital | Hospital Hook-up First, Then Home Hook-up
Started | 47 | 48
Completed | 47 | 48
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Home Hook-up First Then Hook-up in the Hospital | Hospital Hook-up First, Then Home Hook-up
Started | 47 | 48
Completed | 47 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: patients suspected of OSA
Arm/Group | Polysomnography for Suspicion of SDB
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 102
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 70
Region of Enrollment [Number; unit: participants]
  Belgium | 102

OUTCOME MEASURES:

1. Primary Outcome: Failure Rate of Sleep Study
Description: failure rate of polysomnography according to the hook-up protocol. Polysomnographies scored as "poor" or "unsatisafctory" according to Redline et al. SLEEP 1998 are considered as failed.
Time Frame: 1 day
Measure: Number; unit: percentage of participants
Groups:
- Home Hook up First: adults, suspects of suffering from sleep disordered-breathing, who must undergo a diagnostic polysomnography
  polysomnography: home-based polysomnography with home hook-up first
- Lab Hook up First: adults, suspects of suffering from sleep disordered-breathing, who must undergo a diagnostic polysomnography
  polysomnography:home polysomnography with in-lab hook up first
Arm/Group | Home Hook up First | Lab Hook up First
Number analyzed (Participants) | 47 | 48
percentage of participants | 6 | 6

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Home Hook up First: adults, suspects of suffering from sleep disordered-breathing, who must undergo a diagnostic polysomnography
  polysomnography: home-based polysomnography with hook-up performed at home
- Lab Hook up First: adults, suspects of suffering from sleep disordered-breathing, who must undergo a diagnostic polysomnography
  polysomnography: home-based polysomnography with hook-up performed in the sleep lab
Arm/Group | Home Hook up First | Lab Hook up First
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/48
Other Adverse Events (participants affected / at risk) | 0/51 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes